CLINICAL TRIAL: NCT04678206
Title: A Randomized, Adaptive, Double-Blind, Placebo-Controlled, Parallel-Arm, Phase 2b Study to Evaluate the Efficacy and Safety of Multiple Doses of BLU-5937 in Adult Participants With Refractory Chronic Cough
Brief Title: Evaluation of the Efficacy and Safety of BLU-5937 in Adults With Refractory Chronic Cough
Acronym: SOOTHE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bellus Health Inc. - a GSK company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BUS-P2-02; 2020-004136-17 (EudraCT Number)
Record Dates: First submitted 2020-12-09; First posted 2020-12-21 (Actual); Last update posted 2021-12-13 (Actual); Status verified 2021-12

CONDITIONS: Refractory Chronic Cough
Keywords: BLU-5937; Refractory Chronic Cough; P2X3 receptor antagonist
MeSH Terms: conditions — Chronic Cough | interventions — BLU-5937

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- BLU-5937 Dose A (Experimental): BLU-5937 oral dose A twice a day.
  Interventions: Drug: BLU-5937
- BLU-5937 Dose B (Experimental): BLU-5937 oral dose B twice a day.
  Interventions: Drug: BLU-5937
- BLU-5937 Dose C (Experimental): BLU-5937 oral dose C twice a day.
  Interventions: Drug: BLU-5937
- Placebo (Placebo Comparator): Matching Placebo for BLU-5937 oral dose twice a day.
  Interventions: Drug: Placebo
- BLU-5937 Dose A (Population with baseline cough < 25 coughs/hour) (Experimental): BLU-5937 oral dose A twice a day.
  Interventions: Drug: BLU-5937
- Placebo (Population with baseline cough < 25 coughs/hour) (Placebo Comparator): Matching Placebo for BLU-5937 oral dose twice a day.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BLU-5937 — Oral administration of BLU-5937 Tablets
  Arms: BLU-5937 Dose A; BLU-5937 Dose A (Population with baseline cough < 25 coughs/hour); BLU-5937 Dose B; BLU-5937 Dose C
Drug: Placebo — Oral administration of matching placebo for BLU-5937 Tablets
  Arms: Placebo; Placebo (Population with baseline cough < 25 coughs/hour)

SUMMARY:
This is a randomized, double-blind, placebo-controlled, parallel-arm, Phase 2b adaptive dose-finding study of BLU-5937 in participants with Refractory Chronic Cough (RCC).

DETAILED DESCRIPTION:
The primary objective of this study is to determine the therapeutic dose of BLU-5937 in patients with refractory chronic cough by assessing the change from baseline to week 4 in the 24-hour cough frequency with BLU-5937 relative to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving signed informed consent
* Refractory chronic cough (including unexplained chronic cough) for at least one year
* Women of child-bearing potential must use a highly effective contraception method during the study and for at least 14 days after the last dose

Exclusion Criteria:

* Current smoker/vaper (all forms of smoking and inhaled substances, including , cannabis/tobacco smoke and nicotine vapors) or individuals who have given up smoking within the past 6 months, or those with >20 pack-year smoking history
* Diagnosis of Chronic Obstructive Pulmonary Disease (COPD), bronchiectasis, idiopathic pulmonary fibrosis or uncontrolled asthma
* Respiratory tract infection within 4 weeks before screening
* Laboratory confirmed Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) infection at screening
* History of malignancy in the last 5 years
* History of alcohol or drug abuse within the last 3 years
* Has a positive serologic test for human immunodeficiency virus (HIV), hepatitis B virus surface antigen, or hepatitis C virus.
* Previous participation in a BLU-5937 trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2020-12-07 (Actual); Primary Completion 2021-10-21 (Actual); Study Completion 2021-11-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the 24-hour cough frequency | Week 4
  Assessed using an ambulatory cough monitor

SECONDARY OUTCOMES:
Percentage of Participants with a Reduction from Baseline in the 24-hour Cough Frequency by ≥ 30%, 50% and 70% | Week 4
  Assessed using an ambulatory cough monitor
Change from Baseline in Leicester Cough Questionnaire (LCQ) | Week 4
  The LCQ is a patient-reported quality of life (QOL) measure of chronic cough. The questionnaire consists of 19 items to which the patient responds on a 7-point Likert response scale (from 1 to 7). Each item assesses symptoms during cough and the effect of cough on 3 main domains: physical, psychological and social. Domain scores range from 1-7, and the total score ranges from 3 - 21; a higher score indicates a better quality of life.
Change from baseline in cough severity | Week 4
  Assessed by Cough Severity Visual Analogue Scale [VAS] by the participant on a 100 mm visual analog scale where higher scores indicate worse severity.
Incidence (% of subjects) of treatment-emergent adverse events (TEAEs) | 2 Weeks after the last study medication intake
Severity (mild, moderate, or severe) of treatment-emergent adverse events (TEAEs) | 2 Weeks after the last study medication intake

CONTACTS AND LOCATIONS:
Locations (116):
- United States (55):
  - Phoenix Medical Research Inc, Peoria, Arizona
  - Little Rock Allergy and Asthma Clinical Research Center, Little Rock, Arkansas
  - Southern California Institute For Respiratory Diseases, Inc, Los Angeles, California
  - Allergy and Asthma Associates of Southern California, Mission Viejo, California
  - California Medical Research Associates, Inc., Northridge, California
  - Allergy Associates Medical Group Inc., San Diego, California
  - Allergy and Asthma Associates of Santa Clara Valley Research Center, San Jose, California
  - Colorado Allergy and Asthma Centers, Denver, Colorado
  - St. Francis Medical Institute, Clearwater, Florida
  - Floridian Clinical Research, Hialeah, Florida
  - Sweet Hope Research Specialty, Inc., Hialeah, Florida
  - Sher Allergy Specialist/Center for Cough, Largo, Florida
  - Medical Research of Central Florida, Leesburg, Florida
  - ProCare Clinical Research, Miami Lakes, Florida
  - Central Florida Pulmonary Group PA, Orlando, Florida
  - Lenus Research & Medical Group, Sweetwater, Florida
  - IACT Health - Columbus, Columbus, Georgia
  - IACT Health - Lawrenceville, Lawrenceville, Georgia
  - IACT Health - Rincon, Rincon, Georgia
  - Sneeze Wheeze and Itch Associates LLC, Normal, Illinois
  - AES - Synexus Clinical Research US, Inc. - Evansville, Evansville, Indiana
  - Abraham Research PLLC, Fort Mitchell, Kentucky
  - Infinity Medical Research Inc, North Dartmouth, Massachusetts
  - Minnesota Lung Center, Edina, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Minnesota Lung Center, Woodbury, Minnesota
  - The Lung Research Center, LLC, Chesterfield, Missouri
  - University of Missouri, ENT and Allergy Center of Missouri, Columbia, Missouri
  - The Clinical Research Center LLC, St Louis, Missouri
  - Montana Medical Research, Missoula, Montana
  - Creighton University Medical Center, Omaha, Nebraska
  - Atlantic Respiratory Institute, Summit, New Jersey
  - Albuquerque Clinical Trials Inc, Albuquerque, New Mexico
  - CHEAR Center LLC, The Bronx, New York
  - American Health Research Inc, Charlotte, North Carolina
  - Clinical Research of Gastonia, Gastonia, North Carolina
  - Southeastern Research Center, Winston-Salem, North Carolina
  - Bernstein Clinical Research Center Inc, Cincinnati, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Remington Davis Inc, Columbus, Ohio
  - Vital Prospects Clinical Research Institute PC, Tulsa, Oklahoma
  - Clinical Research Associates Of Central Pa, Altoona, Pennsylvania
  - Synexus Clinical Research US, Inc., Anderson, South Carolina
  - National Allergy and Asthma Research, Charleston, South Carolina
  - Clinical Research of Rock Hill, Rock Hill, South Carolina
  - Clinical Trials Center of Middle Tennessee, Franklin, Tennessee
  - Pharmaceutical Research & Consulting Inc, Dallas, Texas
  - El Paso Pulmonary Association, El Paso, Texas
  - Village Research, LLC, Houston, Texas
  - Metroplex Pulmonary and Sleep Medicine Center, McKinney, Texas
  - Diagnostics Research Group, San Antonio, Texas
  - Sherman Clinical Research, Sherman, Texas
  - Allergy Asthma Research Institute, Waco, Texas
  - Intermountain Clinical Research, Draper, Utah
  - TPMG Lung & Sleep Specialist, Williamsburg, Virginia
- Canada (6):
  - McMaster University Medical Centre, Hamilton, Ontario
  - Diex Recherche - Québec, Québec, Quebec
  - Clinique Spécialisée en Allergie de la Capitale, Québec, Quebec
  - Inspiration Research Limited, Toronto, Quebec
  - C I C Maurice Inc, Trois-Rivières, Quebec
  - Diex Recherche - Victoriaville, Victoriaville, Quebec
- Czechia (7):
  - MUDr. I. Cierná Peterová s.r.o., Brandýs nad Labem-Stará Boleslav, Central Bohemia
  - Pneumologie Varnsdorf S.r.o., Nový Bor, Liberec
  - Plicní ambulance Rokycany s.r.o., Rokycany, Plzeň
  - Synexus Czech s.r.o., Prague, Prague
  - MediTrial s.r.o., Jindřichův Hradec, South Bohemia
  - MUDr. Jaroslav Mares - odborny lekar pro obor tuberkulosa a respiracni nemoci, Strakonice, South Bohemia
  - Plicni stredisko Teplice s.r.o., Teplice, Ústí Nad Labem
- Germany (10):
  - Thoraxklinik-Heidelberg gGmbH, Heidelberg, Baden-Wurttemberg
  - Synexus Frankfurt Research Centre, Frankfurt am Main, Hesse
  - IKF Pneumologie, Frankfurt am Main, Hesse
  - Zentrum für ambulante pneumologische Forschung Marburg GbR, Marburg, Hesse
  - Ballenberger. Freytag. Wenisch - Institut fuer klinische Forschung GmbH, Neu-Isenburg, Hesse
  - Kfns Klinische Forschung Schwerin, Schwerin, Mecklenburg-Vorpommern
  - Universitätsklinikum Bonn, Bonn, North Rhine-Westphalia
  - Klinische Forschung Dresden GmbH (KFGN), Dresden, Saxony
  - Synexus Leipzig Research Centre, Leipzig, Saxony
  - Ärztezentrum Axel Springer Passage, Berlin
- Hungary (6):
  - Da Vinci Maganklinika, Pécs, Baranya
  - Synexus Gyula - Magyarország Egészségügyi Szolgáltató Kft, Gyula, Bekes County
  - Dr. Kenessey Albert Korhaz-Rendelointezet, Balassagyarmat, Nógrád megye
  - Szent Borbála Kórház, Tatabánya, Nógrád megye
  - Synexus Zalaegerszeg Magyarország Egészségügyi Kft, Zalaegerszeg, Zala County
  - Synexus Budapest - Magyarország Egészségügyi Szolgáltató Kft, Budapest
- Poland (14):
  - Osrodek Badan Klinicznych CLINSANTE S.C. Ewa Galczak-Nowak Malgorzata Trzaska, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Medical Center Kermed, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Centrum Medyczne Bydgoszcz - PRATIA, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Alergo-Med Specjalistyczna Przychodnia Lekarska Sp. z.o.o, Tarnów, Lesser Poland Voivodeship
  - KLIMED, Bychawa, Lublin Voivodeship
  - Clinical Best Solutions -Lublin, Lublin, Lublin Voivodeship
  - Centrum Alergologii Specjalistyczna Przychodnia Alergologiczna, Lublin, Lublin Voivodeship
  - Centrum Medyczne Warszawa - PRATIA, Warsaw, Masovian Voivodeship
  - Prywatny Gabinet Internistyczno-Alergologiczny, Bialystok, Podlaskie Voivodeship
  - Synexus Polska Sp. z o.o. Oddzial w Gdansku, Gdansk, Pomeranian Voivodeship
  - Synexus Polska Sp. z o.o. Oddzial w Czestochowie, Częstochowa, Silesian Voivodeship
  - Centrum Medyczne Wos i Piwowarczyk, Kraków, Łódź Voivodeship
  - Synexus Polska Sp. Z o.o Oddzial w Lodzi, Lodz, Łódź Voivodeship
  - Ostrowieckie Centrum Medyczne Spólka Cywilna Anna Olech-Cudzik, Krzysztof Cudzik, Ostrowiec Świętokrzyski, Świętokrzyskie Voivodeship
- United Kingdom (18):
  - Synexus Midlands Clinical Research Centre, Birmingham, England
  - West Walk Surgery, Bristol, England
  - MeDiNova Northamptonshire Quality Research Site, Corby, England
  - Castle Hill Hospital, Cottingham, England
  - MeDiNova Warwickshire Quality Research Site, Kenilworth, England
  - Kings College Hospital, London, England
  - Royal Brompton Hospital, London, England
  - NW Consortium Manchester, Manchester, England
  - Wythenshawe Hospital - PPDS, Manchester, England
  - MeDiNova North London Quality Research Site, Middlesex, England
  - North Tyneside General Hospital, North Shields, England
  - MeDiNova East London Quality Research Site, Romford, England
  - MeDiNova Yorkshire Quality Research Site, Shipley, England
  - MeDiNova South London Quality Research Site, Sidcup, England
  - MeDiNova West London Quality Research Site, Wokingham, England
  - Ormeau Clinical Trials Limited, Belfast, Northern Ireland
  - Belfast City Hospital, Belfast, Northern Ireland
  - AES - Synexus Scotland Clinical Research Centre, Glasgow, Scotland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Smith JA, Birring SS, Blaiss MS, McGarvey L, Morice AH, Sher M, Carroll KJ, Garin M, Lanouette S, Shaw J, Yang R, Bonuccelli CM. Camlipixant in Refractory Chronic Cough: A Phase 2b, Randomized, Placebo-controlled Trial (SOOTHE). Am J Respir Crit Care Med. 2025 Jun;211(6):1038-1048. doi: 10.1164/rccm.202409-1752OC. PMID 40043302